CLINICAL TRIAL: NCT06360679
Title: Clinical Feasibility Study of the BariTon™ System in Obese or Overweight (BMI > 27) Patients
Brief Title: Clinical Feasibility Study of the BariTon™ System in Obese or Overweight Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BariaTek Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP000004
Record Dates: First submitted 2024-03-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BariTon™ System implantation (Experimental)
  Interventions: Device: Endoscopic gastric restriction and biliodigestive diversion

INTERVENTIONS:
Device: Endoscopic gastric restriction and biliodigestive diversion — The BariTon™ is endoscopically implanted and retrieved once treatment is completed

SUMMARY:
Safety and efficacy evaluation of the BariTon™, BariaTek Medical gastric restriction and biliodigestive diversion device.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 25 and 60 years inclusive
2. A BMI between 30.0 and 40.0 kg/m2 inclusive with a history of obesity for at least 2 years and a history of failure of supervised weight loss program
3. Stable weight, i.e. < 5% change in body weight for minimum of 3 months prior to enrolment
4. Willing and able to provide written informed consent
5. Willing and able to comply with the study procedures and follow-up schedule

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the BariTon™ | 3 months
  Number of patients with device implantation procedure success
Safety of the BariTon™ | 3 months
  Incidence of device related adverse events

SECONDARY OUTCOMES:
Safety of the BariTon™ | 1 year
  Number of patients with device retrieval procedure success
Safety of the BariTon™ | 1 year
  Incidence of device related adverse events
Efficacy of the BariTon™ | 1 year
  Assessment of clinical variables and other metrics (exploratory)
Efficacy of the BariTon™ | 1 year
  Changes and number of diabetes medication taken
Efficacy of the BariTon™ | 1 year
  Changes and number of statins medication taken
Efficacy of the BariTon™ | 1 year
  Changes and number of blood pressure lowering medication taken
Efficacy of the BariTon™ | 1 year
  Score changes in Weight related Quality of Life using IWQOL-Lite Questionnaire
Efficacy of the BariTon™ | 1 year
  Score changes in food craving using CoEQ Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Sartoretto, Dr, Principal Investigator — The BMI Clinic
Locations (2):
- Australia (2):
  - BMI Clinic Double Bay, Sydney, New South Wales
  - BMI Clinic Liverpool, Sydney, New South Wales